CLINICAL TRIAL: NCT00936806
Title: Observational Study of the Differences in Characteristics of the Spontaneous Electroencephalogram, Derived From the Left and Right Hemisphere in Patients With Unilateral Intracranial Tumor During Routine Anesthesia. Comparison With a Control Group Without Intracranial Pathology.
Brief Title: Observational Study of the Differences in Characteristics of the Spontaneous Electroencephalogram, Derived From the Left and Right Hemisphere in Patients With Unilateral Intracranial Tumor During Routine Anesthesia: Comparison With a Control Group Without Intracranial Pathology
Acronym: VISTA
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2008/666
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Intracranial Tumor
Keywords: Intracranial tumor patients
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Unilateral intracranial tumor: Subjects with unilateral intracranial tumor
- Control group: Subjects without intracranial pathology

SUMMARY:
Study of the influence of brain tumor on bilateral electroencephalogram (EEG) during anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 - 80 years old
* Able to comprehend, sign, and date the written informed consent document to participate in the clinical trial
* Scheduled for "procedure"
* ASA Class I, II or III as assigned by the anaesthesiologist

Exclusion Criteria:

* Allergy or inability to tolerate "product"
* Body weight less than 70% or more than 130% of ideal body weight
* Pregnant or nursing females
* Participation in a clinical trial within the past 30 days
* Congenital mental disability or congenital anatomical brain abnormality
* A medical history of cerebrovascular accident or thrombosis
* A medical history of carotic artery occlusive pathology
* A medical history of degenerative cerebral pathology (MS, Dementia, ALS, para-or tetraplegia due to a traumatic disruption of the spinal cord)
* A medical history of severe psychiatric pathology (Schizophrenia, severe depression, alcoholism, drug abuse) Mild depression evoked by coping with the diagnosis of cancer is not excluded
* Patients with a history of epileptic insults. Patients receiving preventive anti-epileptic treatment due to the tumoral process are not excluded.
* Patients with low cardiac output conditions due to pre-existing cardiac pathology (Cardiac insufficiency, valve pathology, dysrhythmia, myocardial infarction). Patients presenting with stable coronary artery disease with a normal myocardial function are not excluded)
* Arterial hypertension is not an exclusion criteria, nor is the use of antihypertensive medication, except beta blockers for their potential interfering effects on spontaneous EEG.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unilateral intracranial tumor during routine anesthesia at the University Hospital Ghent
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Asymmetry of EEG extracted indices obtained from either healthy or diseased hemispheres. | 2 years

SECONDARY OUTCOMES:
Covariates that causes asymmetry between bilaterally derived EEG. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Vereecke, MD PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website of the University Hospital Ghent — http://www.uzgent.be